CLINICAL TRIAL: NCT05652686
Title: An Open-label, Multicenter, Dose Escalation, and Dose Expansion Phase 1/2 Study With Peluntamig (PT217) Followed by a Key ChemotherapY and/or Checkpoint Inhibitor ComBination in Patients With NeuRoendocrIne Carcinomas That Are Known to be DLL3 expressinG CancErs (SKYBRIDGE)
Brief Title: A Study of Peluntamig (PT217) in Patients With Neuroendocrine Carcinomas Expressing DLL3 (the SKYBRIDGE Study)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Phanes Therapeutics (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PT217X1101
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Small Cell Lung Cancer (SCLC); Large Cell Neuroendocrine Cancer (LCNEC); Neuroendocrine Prostate Cancer (NEPC); Gastroenteropancreatic Neuroendocrine Carcinoma (GEP-NEC); Neuroendocrine Carcinomas (NEC); Extrapulmonary Neuroendocrine Carcinoma (EP-NEC)
Keywords: DLL3; DLL3 expressing tumors; Lung cancer; SCLC; LCNEC; NEPC; GEP-NEC; Small Cell Lung Cancer; Large cell neuroendocrine cancer; Neuroendocrine prostate cancer; Gastroenteropancreatic neuroendocrine carcinoma; Neuroendocrine carcinoma; Extrapulmonary neuroendocrine carcinoma; EP-NEC; CD47
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine; Lung Neoplasms | interventions — EC regimen; Paclitaxel; atezolizumab

STUDY DESIGN:
Intervention Model Description: The study will consist of 4 parts: Dose Escalation (Part A), Dose Expansion (Part B), Chemo Combination Therapy (Part C) and ICI combination Therapy (Part D).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A: Dose Escalation (Experimental): A standard 3+3 dose escalation design will be employed.
  Interventions: Drug: Peluntamig (PT217)
- Part B: Dose Expansion (Experimental): Part B cohorts will open after the dose level considered for RDE has been cleared in Parts A, C and D.
  Interventions: Drug: Peluntamig (PT217)
- Part C: Chemotherapy Combination Therapy (Experimental): Part C of the study will include Cohorts C1 and C2, combining Peluntamig (PT217) with chemotherapy.
  Interventions: Drug: Peluntamig (PT217); Drug: Carboplatin + Etoposide; Drug: Paclitaxel.
- Part D: ICI Combination Therapy (Experimental): In part D, Peluntamig (PT217) will be given in combination with atezolizumab, either alone or in combination with chemotherapy.
  Interventions: Drug: Peluntamig (PT217); Drug: Carboplatin + Etoposide; Drug: Atezolizumab

INTERVENTIONS:
Drug: Peluntamig (PT217) — A bispecific antibody (bsAb) against DLL3 and CD47.
Drug: Carboplatin + Etoposide — Administered per Standard of Care.
  Arms: Part C: Chemotherapy Combination Therapy; Part D: ICI Combination Therapy
Drug: Paclitaxel. — Administered per Standard of Care.
  Arms: Part C: Chemotherapy Combination Therapy
Drug: Atezolizumab — Administered per Standard of Care.
  Arms: Part D: ICI Combination Therapy

SUMMARY:
This is a first-in-human, Phase 1/2, open-label, dose escalation, dose expansion and combination study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of Peluntamig (PT217) as a monotherapy and in combination with chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria

1. NECs that have transformed from NSCLC are not eligible. Part A: Patients with histologically or cytologically confirmed unresectable advanced or metastatic small cell lung cancer (SCLC), large cell neuroendocrine carcinoma of the lung (LCNEC), or extrapulmonary neuroendocrine carcinoma (EP-NEC). Patients with tumors that are of mixed histology are eligible only if neuroendocrine carcinoma/small cell cancer component is predominant and represents at least 50% of the overall tumor tissue. Patients with well differentiated grade 3 neuroendocrine tumors (Ki-67 ≥ 55%) may be considered if their tumors are DLL3 positive.

   Patients may have progressed after standard of care treatments (at least one line of platinum-based chemotherapy with or without immune checkpoint inhibitor for SCLC patients) or other treatment options, or for whom treatment is not available or not tolerated.

   Part B: Patients must meet the same criteria in Part A, C or D.

   Part C:

   • Cohort C1: patients with LCNEC or EP-NEC eligible for first-line (1L) CE treatment. SCLC patients who have relapsed on a 1L treatment (including platinum-based therapy with or without ICI) but remain platinum sensitive (defined as patients who experienced disease progression at least 90 days after their last platinum based chemotherapy) and are eligible for CE treatment rechallenge.

   Cohort C2: patients with SCLC, LCNEC and EP-NEC eligible for second line (2L) paclitaxel treatment.

   Part D:
   * Cohort D1: will include 2L patients with SCLC, LCNEC, pr EP-NEC that have progressed/relapsed from their first-line treatment that may have included an ICI.
   * Cohort D2: will include 1L ES-SCLC patients that have completed their induction therapy with carboplatin and etoposide plus atezolizumab and are eligible to continue with atezolizumab. These patients must have either stable disease or partial response prior to enrollment.
   * Cohort D3: will include 1L ES-SCLC patients that are treatment naïve or have received C1D1/2/3 and are eligible for treatment with CE plus atezolizumab.
2. Able to provide a formalin fixed, paraffin embedded (FFPE) tumor tissue sample (preferably a newly acquired biopsy, or if not possible, archival tissue) to be assessed for DLL3 expression and other biomarkers.
3. ECOG performance status of 0 or 1.
4. Adequate organ function confirmed at screening and within 72 hours of initiating C1D1 of Peluntamig (PT217) treatment.

Key Exclusion Criteria

1. Women who are pregnant or lactating.
2. Women of child-bearing potential (WOCBP) who do not use adequate birth control.
3. Autoimmune disease requiring systemic treatment within the past twelve months.
4. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2, and excluding ICIs) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment with Peluntamig (PT217).
5. Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications (≥ 10 mg prednisone, or equivalent) within 14 days prior to study drug Peluntamig (PT217), or anticipation of need for systemic immunosuppressive medication during study drug Peluntamig (PT217).
6. Patients who have experienced Grade ≥ 3 immune-related events, such as (non-infectious) pneumonitis, interstitial lung disease, myocarditis.
7. Treatment with therapeutic oral or i.v. antibiotics within 2 weeks prior to initiation of study treatment with Peluntamig (PT217).
8. Patients with untreated brain or central nervous system (CNS) metastases or brain/CNS metastases that have progressed.

   Note: Patients with treated brain metastases that are off corticosteroids and have been clinically stable for 14 days are eligible for treatment.
9. Impaired cardiac function or significant diseases.
10. For Part D only, uncontrolled hypercalcemia.
11. For Part D only, significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
12. Prior hemolytic anemia or Evans Syndrome in the last 3 months.
13. Patients who have Grade ≥ 3 neuropathy.
14. Patients who are currently receiving treatment with therapeutic doses of warfarin sodium (Coumadin®) or any other coumarin-derivative anticoagulants .

Additional criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
To determine the dose-limiting toxicity (DLT) of Peluntamig (PT217). | Through study completion.
To determine the maximum tolerated dose (MTD) of Peluntamig (PT217) if reached. | Through study completion.
To determine recommended dose for expansion (RDE) of Peluntamig (PT217). | Through study completion.
To evaluate the safety and tolerability of Peluntamig (PT217). | Through study completion.
To evaluate the efficacy of Peluntamig (PT217) monotherapy or in combination treatments | Through study completion

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of Peluntamig (PT217). | Through study completion.
To evaluate the immunogenicity (ADA) of Peluntamig (PT217). | Through study completion.
To further evaluate the efficacy of Peluntamig (PT217) monotherapy or in combination treatments | Through study completion.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine (Siteman Cancer Center), St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Sarah Cannon Research Institute University of Oklahoma, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Mays Cancer Center / University of Texas, San Antonio, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided